CLINICAL TRIAL: NCT05509634
Title: Compared With Fosaprepitant Dimeglumine for Injection and Palonosetron Hydrochloride Injection, to Evaluate the Efficacy and Safety of HR20013 for Injection for Prevention of Chemotherapy-induced Nausea and Vomiting After Highly Emetogenic Chemotherapy
Brief Title: Clinical Study of HR20013 for Injection in Patients With Malignant Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HR20013-301
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-09

CONDITIONS: Prevention of Nausea and Vomiting Caused by Highly Emetogenic Chemotherapy
MeSH Terms: interventions — fosaprepitant

STUDY DESIGN:
Intervention Model Description: HR20013 for injection + dexamethasone compared with fosaprepitant dimeglumine for injection + palonosetron hydrochloride injection + dexamethasone
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): HR20013 for injection + simulant of fosaprepitant dimeglumine for injection + simulant of palonosetron hydrochloride injection + dexamethasone
  Interventions: Drug: HR20013 for injection；dexamethasone
- Treatment group B (Active Comparator): simulant of HR20013 for injection + fosaprepitant dimeglumine for injection + palonosetron hydrochloride injection + dexamethasone + simulant of dexamethasone
  Interventions: Drug: fosaprepitant dimeglumine for injection；palonosetron hydrochloride injection；dexamethasone

INTERVENTIONS:
Drug: HR20013 for injection；dexamethasone — HR20013 for injection；Drug for preventing nausea and vomiting caused by chemotherapy
  dexamethasone: Drug for preventing nausea and vomiting caused by chemotherapy
  Arms: Treatment group A
Drug: fosaprepitant dimeglumine for injection；palonosetron hydrochloride injection；dexamethasone — fosaprepitant dimeglumine for injection: Drug for preventing nausea and vomiting caused by chemotherapy
  palonosetron hydrochloride injection: Drug for preventing nausea and vomiting caused by chemotherapy
  dexamethasone: Drug for preventing nausea and vomiting caused by chemotherapy
  Arms: Treatment group B

SUMMARY:
To evaluate the efficacy and safety of HR20013 for injection for prevention of chemotherapy-induced nausea and vomiting after highly emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, of either gender
2. Has a diagnosed malignant tumor
3. has never been treated with chemotherapy and is to receive the first course of cisplatin-based chemotherapy
4. Predicted life expectancy of ≥ 3 months
5. Has a performance status (ECOG scale) of 0 to 1
6. Adequate bone marrow, kidney, and liver function
7. Women of childbearing potential must have negative pregnancy test (serum test) results within 72 hours prior to enrollment
8. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Scheduled to receive any radiation therapy to the abdomen or pelvis from Day -7 through Day 8
2. Scheduled to receive any other chemotherapeutic agent with an high emetogenicity level from Day 2 through Day 8
3. Has taken the following agents within the last 48 hours 5-HT3 antagonists, Phenothiazines, Benzamides, Domperidone, Cannabinoids, Benzodiazepines
4. Subjects receiving palonosetron hydrochloride within 14 days before randomization
5. Subjects who previously received NK-1 receptor antagonists within 28 days prior to randomization
6. Subjects with a history of myocardial infarction or unstable angina pectoris
7. Subjects with atrioventricular block or cardiac insufficiency
8. Subjects with poor blood pressure control after medication
9. Subjects with symptomatic brain metastases or any symptoms suggestive of brain metastasis or intracranial hypertension
10. Subjects who have experienced emetic events (vomiting or dry vomiting) or nausea within 24 hours before randomization
11. Participated in clinical trials of other drugs (received experimental drugs)
12. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Complete response during the overall phase after the start of the first cisplatin administration | 0-120 hours after the start of the first cisplatin administration
  To compare the rate of subjects achieving and maintaining a complete response (defined as no emetic episode and no need for rescue medication) after the start of the first cisplatin administration.

SECONDARY OUTCOMES:
Complete response during the acute phase, the delayed phase, >120-168 hours, and 0-168 hours after the start of the first cisplatin administration | the acute phase (0-24 hours), the delayed phase (>24-120 hours), >120-168 hours, and 0-168 hours after the first cisplatin administration
  To compare the proportion of subjects achieving and maintaining a complete response (defined as no emetic episode and no need for rescue medication) during the specified period.
Complete response during the acute phase, the delayed phase, the overall phase, >120-168 hours, and 0-168 hours after the start of the second cisplatin administration | the acute phase (0-24 hours), the delayed phase (>24-120 hours), the overall phase (0-120 hours), >120-168 hours, and 0-168 hours after the start of the second cisplatin administration
  To compare the proportion of subjects achieving and maintaining a complete response (defined as no emetic episode and no need for rescue medication) during the specified period.
No significant nausea | the acute phase (0-24 hours), the delayed phase (>24-120 hours), the overall phase (0-120 hours), >120-168 hours and 0-168 hours after the start of each cisplatin administration
  To compare the proportion of subjects with no significant nausea (defined as maximum nausea on a visual analogue scale <25 mm) during the specified period.
No nausea | the acute phase (0-24 hours), the delayed phase (>24-120 hours), the overall phase (0-120 hours), >120-168 hours and 0-168 hours after the start of each cisplatin administration
  To compare the proportion of subjects with no nausea (defined as maximum nausea on a visual analogue scale <5 mm) during the specified period.
No emetic | the acute phase (0-24 hours), the delayed phase (>24-120 hours), the overall phase (0-120 hours), >120-168 hours and 0-168 hours after the start of each cisplatin administration
  To compare the proportion of subjects with no emetic event during the specified period.
No rescue medication | the acute phase (0-24 hours), the delayed phase (>24-120 hours), the overall phase (0-120 hours), >120-168 hours and 0-168 hours after the start of each cisplatin administration
  To compare the proportion of subjects who received no rescue medication during the specified period.
Complete protection | the acute phase (0-24 hours), the delayed phase (>24-120 hours), the overall phase (0-120 hours), >120-168 hours and 0-168 hours after the start of each cisplatin administration
  To compare the proportion of subjects with complete protection (defined as patients who experienced no emetic event and received no rescue medication and had no significant nausea) during the specified period).
Total control | the acute phase (0-24 hours), the delayed phase (>24-120 hours), the overall phase (0-120 hours), >120-168 hours and 0-168 hours after the start of each cisplatin administration
  To compare the proportion of subjects with total control (defined as patients who experienced no emetic events and received no rescue medication and had no nausea) during the specified period.
Time to treatment failure | During 0-168 hours after the start of each cisplatin administration
  Time to the first occurrence of emetic event or the first rescue medication.
The score using the functional living index-emesis (FLIE) questionnaire | During 0-168 hours after the start of each cisplatin administration
  To compare the change of score using FLIE questionnaire before and after treatment.
Number of participants with injection site reaction and with treatment-related adverse events as assessed by CTCAE v5.0 | 0 to 504 hours after the start of each cisplatin administration
  To compare the number of participants with injection site reaction and with treatment-related adverse events as assessed by CTCAE v5.0.
plasma concentration of HR20013 | Evaluation time points include 1-2 hours, 5-10 hours, and 3 days after the start of the first HR20013 administration, and day 1 of the second HR20013 administration
  To analyse the plasma concentration of HR20013 at the specified time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center Yuexiu Campus, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou H, Zhao Y, Zhang M, Yao J, Leng S, Li X, Lin L, Chen J, Zhang S, Qin X, Qin Z, Yi T, Wang R, Li X, Yu Y, Wang Z, Zheng Q, Mei J, Zang A, Li N, Cao F, Cao K, Li W, Lu Y, Lin D, Zhou Y, Yang R, Fang W, Zhou N, Yang Y, Zhang Y, Chen G, Zhou T, Yang X, Wang H, Wang Y, Huang Y, Zhang L. Randomized, Phase III Trial of Mixed Formulation of Fosrolapitant and Palonosetron (HR20013) in Preventing Cisplatin-Based Highly Emetogenic Chemotherapy-Induced Nausea and Vomiting: PROFIT. J Clin Oncol. 2025 Mar 20;43(9):1123-1136. doi: 10.1200/JCO-24-01308. Epub 2024 Dec 2. PMID 39621965